CLINICAL TRIAL: NCT04690647
Title: The Efficacy of Ultrasound Guided Suprainguinal Fascia Iliaca Compartment Block for Acute Paint Control After Elective Total Hip Replacement Using Postero-lateral Approach
Brief Title: The Efficacy of Suprainguinal Fascia Iliaca Compartment Block for Analgesia After Elective Total Hip Replacement.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Saint Lucas Hospital, Poland (Other)
Responsible Party: Principal Investigator, Wojciech Gola, MD, Head of The Department of Anesthesia, Saint Lucas Hospital, Poland
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: FasiaIliaca
Record Dates: First submitted 2020-06-04; First posted 2020-12-31 (Actual); Last update posted 2020-12-31 (Actual); Status verified 2020-12

CONDITIONS: Anesthesia, Local; Analgesia; Arthropathy of Hip
MeSH Terms: conditions — Agnosia | interventions — Analgesics, Opioid; Dexamethasone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Opioid and non opioid postoperative analgesia. (Placebo Comparator): Group of patients with opioid and non opioid based postoperative analgesia without preoperative regional anaesthesia and dexamethasone.
  Interventions: Other: Opioid and non opioid postoperative analgesia.
- Regional anaesthesia, opioid and non opioid postoperative analgesia. (Experimental): Group of patients with opioid and non opioid based postoperative analgesia with preoperative regional anaesthesia and without preoperative dexamethasone.
  Interventions: Other: Opioid and non opioid postoperative analgesia.; Other: Fascia iliaca compartment block
- Regional anaesthesia, dexamethasone, opioid and non opioid postoperative analgesia (Experimental): Group of patients with opioid and non opioid based postoperative analgesia with preoperative regional anaesthesia and dexamethasone.
  Interventions: Other: Opioid and non opioid postoperative analgesia.; Other: Fascia iliaca compartment block; Drug: Dexamethasone

INTERVENTIONS:
Other: Opioid and non opioid postoperative analgesia. — Postoperative analgesia will be based on opioid and non opioid analgesics according to standardised protocol.
Other: Fascia iliaca compartment block — Ultrasound guided suprainguinal fascia iliaca compartment block will be performed using 0.375% ropivacaine and 5ug/ml adrenaline according to standardised protocol.
  Arms: Regional anaesthesia, dexamethasone, opioid and non opioid postoperative analgesia; Regional anaesthesia, opioid and non opioid postoperative analgesia.
Drug: Dexamethasone — Dexamethasone will be administered preoperatively in a dose of 0,1 mg/kg.
  Arms: Regional anaesthesia, dexamethasone, opioid and non opioid postoperative analgesia

SUMMARY:
Total hip replacement surgery is one of the most common orthopedic interventions. Proper anaesthesia and adequate analgesia is one of the key interests of attending anaesthetist. Recent studies show that ultrasound guided suprainguinal fascia iliaca compartment block may play a significant role in proper management of pain after these procedures. The aim of this study was to assess the clinical usefulness and compare different methods of anaesthesia for total hip replacement surgery via posterolateral approach.

ELIGIBILITY:
Inclusion Criteria:

* age 18-75 years old
* informed consent to participate in the study
* ASA score I-III
* BMI -19-30kg/m2
* qualified for total hip replacement
* no contraindication to used anesthesia and drugs

Exclusion Criteria:

* contraindications to spinal anesthesia and regional blocks
* previously coexisting chronic pain
* previously opioids intake
* BMI>30kg/m2
* allergy to drugs using during study
* mental status preventing the usage of patient controlled analgesia pump

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2018-09-28 (Actual); Primary Completion 2019-12-20 (Actual); Study Completion 2019-12-20 (Actual)

PRIMARY OUTCOMES:
Opioid consumption [mg] | 48 hours
  Postoperative opioid consumption was noted.
Opioid related adverse effects | 48 hours
  Postoperative incidence of nausea, vomiting, constipation and apnea were noted.
Hospital stay [days] | 31 days
  Total length of hospital stay was noted.

SECONDARY OUTCOMES:
Likert scale | 31 days
  Likert scale value was noted at the discharge. Value of 1 corresponded with strong dissatisfaction, value of 2 with dissatisfaction, value of 3 with neither satisfaction nor dissatisfaction, value of 4 with satisfaction, value of 5 with strong satisfaction.

CONTACTS AND LOCATIONS:
Overall Officials: Wojciech Gola, MD, Principal Investigator — Head of the Department of Anesthesia and Intensive Care Unit, Saint Lucas Hospital, Konskie, Poland
Locations (1):
- Saint Lucas Hospital, Gmina Końskie, Świętokrzyskie Voivodeship, Poland

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Gola W, Bialka S, Owczarek AJ, Misiolek H. Effectiveness of Fascia Iliaca Compartment Block after Elective Total Hip Replacement: A Prospective, Randomized, Controlled Study. Int J Environ Res Public Health. 2021 May 4;18(9):4891. doi: 10.3390/ijerph18094891. PMID 34064427